CLINICAL TRIAL: NCT06375447
Title: Study on an Intelligent Model for the Diagnosis and Treatment of Insomnia Disorder
Brief Title: Intelligent Diagnosis and Treatment Model for Insomnia Disorder
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: West China Hospital (Other); Beijing Tiantan Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Chifeng City Center Hospital Ningcheng County (Unknown)
Responsible Party: Sponsor
Other Study IDs: Insomnia
Record Dates: First submitted 2024-01-01; First posted 2024-04-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Insomnia
Keywords: Insomnia; Intelligence Model; Prediction; Differential diagnosis and treatment; System
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected. The buffy coat of blood collected in an EDTA-tube to obtain plasma, will be stored for the isolation of DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with insomnia: Patients with a complaint about insomnia.
  Interventions: Other: Routine clinical treatment

INTERVENTIONS:
Other: Routine clinical treatment — Routine clinical treatment is based on the latest international guidelines for insomnia.

SUMMARY:
To establish a multicenter, multi-dimensional cohort on insomnia disorder and to develop an intelligent model for the diagnosis and treatment of insomnia disorder.

DETAILED DESCRIPTION:
The study endeavors to establish a multicenter cohort comprising 16,000 individuals diagnosed with insomnia disorder, with a subsequent 2-year follow-up. Objectives encompass elucidating the natural development of insomnia disorder within diverse populations, identifying associated factors, and evaluating the short-term and long-term impacts on physiological, psychological, and social functions in insomnia disorder. Additionally, the research aims to devise early screening methodologies, precise assessments, and innovative disease classifications utilizing real-time assessment technology within the insomnia disorder cohort. Furthermore, the investigation seeks to ascertain graded diagnoses, treatment modalities, and prognostic indicators based on advanced multi-dimensional real-time assessment technology applied to a substantial insomnia disorder cohort. Finally, the study aims to refine remote interactive diagnostic and treatment modalities tailored to diverse age groups, culminating in developing a systematic graded diagnostic and treatment framework for insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

1. A complaint of insomnia;
2. Age between 18 and 75;
3. Able to fill out the scale on their own;
4. Agree to sign the informed consent to participate in the study and cooperate in completing the follow-up visit.

Exclusion Criteria:

1.A current or history of comorbid Axis I psychiatric disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a complaint about insomnia.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of Pittsburgh Sleep Quality Index (PSQI) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.

SECONDARY OUTCOMES:
The change of Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The DBAS assessing sleep related cognitions in 16 item rated on a 10-point Likert scale, and the total score ranges from 0 to 160 with higher scores indicating more intensive disfunctional beliefs.
The change of Epworth Sleepiness Scale (ESS) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The ESS assessing daytime sleepiness consists of 8-items on a 4-point Likert scale, and the total score ranges from 0 to 24 with higher scores indicating more sleepiness.
The change of sleep onset latency from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  Sleep onset latency is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer sleep onset latency).
The change of wake after sleep onset from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  Wake after sleep onset is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer wake after sleep onset).
The change of terminal wakefulness from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  Terminal wakefulness is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer terminal wakefulness).
The change of sleep efficiency from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  Sleep efficiency is assessed with the Carney (2012) consensus sleep diary. This is measured in percentage (higher scores indicating better sleep efficiency).
The change of total sleep time from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  Total sleep time is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer total sleep time).
The change of time in bed from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  Time in bed is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer time in bed).
The change of Insomnia severity index (ISI) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The ISI reporting insomnia symptoms severity consists of 7-items on a 5-point Likert scale, and the total score ranges from 0 to 28 with higher scores indicating more severe insomnia.
The change of Short Form 36 (SF-36) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The SF-36 quantifing the quality of life in relation to health status consists of 36-items with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The total score ranges from 0-100 (the worst possible to the most possible).
The change of PHQ-15 total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The PHQ-15 measuring somatic distress consists of 15 items, and the total score ranges from 0 to 30 with higher scores indicating more severe somatic distress.
The change of PDQ-D-5 total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The PDQ-D-5 assessing perceived cognitive deficits from the patient's perspective consists of 5 items, and the total score ranges from 0 to 20 with higher scores indicating greater perceived deficit.
The change of SHAPS total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The SHAPS assessing anhedonia consists of 14 items, and the total score ranges from 14 to 56 with higher scores indicating more serious the anhedonia.
The change of Life Events Scale (LES) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  The LES assessing the perceived stress and number of stressful life events experienced consists of 48 items which are classified into three dimensions: family life events (28 items), work and study events (13 items), and social events (7 items) with higher scores in LES perceived greater stressfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Wang, MD & PhD, Study Director — Xuanwu Hospital, Beijing
Locations (5):
- China (5):
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital of Soochow University, Suzhou

IPD SHARING:
Plan to Share IPD: No